CLINICAL TRIAL: NCT00549185
Title: An Open-label Multi-dose-escalation, Safety and Pharmacokinetic Study of SAR3419 Administered as a Single Agent by Intravenous Infusion Every 3 Weeks in Patients With Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma (NHL)
Brief Title: Multi-dose-escalation Safety and Pharmacokinetic Study of SAR3419 as Single Agent in Relapsed/Refractory B-cell Non Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED6828; NCT00539682 (obsolete NCT alias)
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Lymphoma; Non-Hodgkin
MeSH Terms: conditions — Lymphoma | interventions — coltuximab ravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SAR3419 — Intravenous infusion

SUMMARY:
The primary objective is to determine the maximum tolerated dose of SAR3419 and to characterize the dose limiting toxicity(ies). Secondary objectives are to determine the anti-lymphoma activity, the global safety and the PK profile.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD19-positive non-Hodgkin's B-cell lymphoma, relapsed or refractory after standard treatments, with no curative option with conventional therapy
* ECOG performance status 0 to 2

Exclusion Criteria:

* Burkitt's lymphoma, Lymphoblastic lymphoma, Chronic lymphocytic leukemia (Small lymphocytic lymphoma may be included)
* Chemotherapy or radiation therapy or other investigational agents within 4 weeks prior to entering the study
* Previous radioimmunotherapy within 12 weeks
* Known intolerance to infused protein products or maytansinoids
* Poor kidney, liver and bone marrow functions
* Any serious active disease or co-morbid condition, which in the opinion of the principle investigator, will interfere with the safety or with compliance with the study
* Pregnant or breast-feeding women
* Patient with reproductive potential without effective birth control methods

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicity(ies) at each tested dose level | Study period

SECONDARY OUTCOMES:
Tumor response (complete response, partial response, stable disease) according to Cheson criteria and duration of response | Study period
Incidence of Adverse Events | Study period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States